CLINICAL TRIAL: NCT04556019
Title: Results of the Surgical Treatment of Patients From Hepatobiliopancreatic Surgical Unit at the Complejo Hospitalario de Navarra
Brief Title: Results of Surgical Treatment of the Hepatobiliopancreatic Surgical Unit
Acronym: HPB
Status: Recruiting | Type: Observational
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Other Study IDs: CIRUGIA HPB-CHN
Record Dates: First submitted 2019-06-11; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Pancreas Disease; Liver Diseases; Surgical Procedure, Unspecified; Bile Duct Diseases
Keywords: Hepatobiliopancreatic surgery
MeSH Terms: conditions — Pancreatic Diseases; Liver Diseases; Bile Duct Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hepatobiliopancreatic surgery — Different surgical techniques tailored to each patient´s pathology

SUMMARY:
The main aims of this study are:

1. - to evaluate post-surgical morbidity and mortality outcomes, following the criteria and the definitions from Claven-Dindo and ISGPS international classifications, of the patients operated by the HPB Surgical Unit.
2. - to evaluate survival and disease-free survival rates of the patients operated by the HPB Surgical Unit due to tumoral cause.

ELIGIBILITY:
Inclusion Criteria:

* All patients operated by the HPB Surgical Unit in the last 10 years (retrospective)
* All patients being operated by the HPB Surgical Unit from January 2019 onwards who provide inform consent (prospective).

Exclusion Criteria:

* Patients not eligible for surgery
* Patients not interested in taking part in the study

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All out-patients and in-patients at the HPB Surgical Unit
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patient with post-surgical morbidity and mortality operated by the HPB Surgical Unit | 90 days post-surgery
  Morbidity and mortality outcomes are evaluated following the criteria and definitions from Claven-Dindo and ISGPS international classifications
Survival rate of patients operated by the HPB Surgical Unit | 5-years post-surgery
  These patients are operated due to tumoral cause
Disease-free survival rate of patients operated by the HPB Surgical Unit | 5-years post-surgery
  These patients are operated due to tumoral cause

SECONDARY OUTCOMES:
Assessment of standardization of pre and post-surgical care | 90 days
Evaluation of the result of the multimodal treatment | 90 days
Assessment of the oncological quality standards of patients operated by HPB Surgical Unit due to tumoral cause | 5 years
Assessment of the results from minimally invasive techniques in HPB surgery | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Herrera Cabezón, MD, Principal Investigator — Complejo Hospitalario de Navarra
Locations (1):
- Complejo Hospitalario de Navarra, Pamplona, Navarre, Spain